CLINICAL TRIAL: NCT01209364
Title: Double-Blind, Randomized, Parallel Group, Multicenter Study of Durolane Compared to Methylprednisolone in Subjects With Osteoarthritis of the Knee
Brief Title: Durolane Versus Methylprednisolone in Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 35GA0608
Record Dates: First submitted 2010-09-20; First posted 2010-09-27 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2007-08

CONDITIONS: Knee Osteoarthritis
Keywords: comparative; randomized; double-blind; non-inferior; knee OA
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Durolane (Experimental): intraarticular hyaluronic acid
  Interventions: Device: Durolane is a device, methylprednisolone in a drug
- methylprednisolone (Active Comparator): intraarticular injection
  Interventions: Device: Durolane is a device, methylprednisolone in a drug

INTERVENTIONS:
Device: Durolane is a device, methylprednisolone in a drug — single intraarticular injection
  Other Names: Durolane and Depo-Medrol are the brand names

SUMMARY:
The primary objective is to determine whether Durolane is non-inferior to methylprednisolone, as assessed by level of pain, when each are given as single intra-articular injections for the relief of pain, in the treatment of symptomatic osteoarthritis of the knee at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject (female or male) 35-80 years of age
* Unilateral knee pain
* Radiographic evidence of OA
* WOMAC pain score of 7-17
* Subject normally active
* Subject has attempted but not responded adequately to previous non-pharmacological therapy(ies);
* Subject cooperative and able to communicate effectively with the investigators;
* Body mass index ≤ 40 kg/m2;
* Signed informed consent obtained.

Exclusion Criteria:

* Knee effusion
* Contralateral knee OA
* Clinically significant joint pain from joints other than the knee
* Previous intra-articular steroid injection into the study knee within the last 3 months;
* Previous intra-articular HA injection into the study knee within the last 9 months;
* Previous allergic type reaction to a HA product, a steroid, or lidocaine/related anesthetics;
* Treatment with analgesics other than paracetamol (acetaminophen) (including topical agents for the knee) within 5 half lives of the drug prior to the baseline visit;
* Use of systemic glucocorticosteroids (excluding inhaled steroids) within the last 3 months;
* Treatment with glucosamine/chondroitin sulfate initiated within the past 3 months
* Change in physical therapy for the knee within the last three months
* Arthroscopy or other surgical procedure in the study knee within the past 12 months;
* Any planned arthroscopy or other surgical procedure during the study period;
* Previous history or presence of active septic arthritis
* Active skin disease or infection in the area of the injection site;
* Systemic active inflammatory condition or infection
* Bleeding diathesis or use of anticoagulants
* Current uncontrolled diabetes mellitus;
* Any medical condition that in the opinion of the investigator makes the subject unsuitable for inclusion
* Pregnant or breastfeeding woman or woman of childbearing potential not practicing adequate contraception;
* Involvement in other clinical trials

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2007-03; Primary Completion 2008-01 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Pain level and responder rate | up to 12 weeks

SECONDARY OUTCOMES:
WOMAC stiffness score | 26 weeks blinded phase + 26 weeks OLE
  Will be assessed at each clinic visit
WOMAC physical function | 26 weeks blinded phase + 26 weeks OLE
  Will be assessed at each clinic visit
Functional assessment | 26 weeks blinded phase + 26 weeks OLE
  Will be assessed at each clinic visit
Safety assessment (Adverse Events) | 26 weeks blinded phase + 26 weeks OLE
  Will be assessed at each clinic visit using standard questions

CONTACTS AND LOCATIONS:
Locations (23):
- Canada (15):
  - Alberta Bone & Joint Health Institute, Calgary, Alberta
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - Orthopaedic & Sport Medicine Institute of Nova Scotia, Halifax, Nova Scotia
  - Dr. Wilson, Lunenburg, Nova Scotia
  - QEII Health Sciences Centre-New Halifax Infirmary, Halifax, Ontario
  - Charlton Medical Centre, Hamilton, Ontario
  - MAC Research Inc., Hamilton, Ontario
  - Fowler Kennedy Sport Medicine Clinic, London, Ontario
  - Credit Valley Rheumatology, Mississauga, Ontario
  - The Arthritis Program Research Group, Newmarket, Ontario
  - Dr. Dobson, Peterborough, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Sport C.A.R.E. Women's College Hospital, Toronto, Ontario
  - Centre de Rhumatologie St-Louis, Saint-Foy, Quebec
  - Saskatoon Osteoporosis Centre, Saskatoon, Saskatchewan
- Sweden (4):
  - Läkargruppen Kristinelund, Gothenburg
  - Ortopediska huset, Johanneshov
  - Läkarhuset Ellenbogen, Malmo
  - Ortopediska huset, Stockholm
- United Kingdom (4):
  - Kings College Hospital - Department of Rheumatology, London
  - Newcastle University Clinical Research FacilityRoyal Victoria Infirmary, Newcastle
  - Robert Jones and Agnes Hunt Orthopaedic & District Hospital - Institute of Orthopaedics, Oswestry
  - Southampton General Hospital - MRC Epidemiology Resource Center, Southampton

REFERENCES:
- [Derived] Leighton R, Akermark C, Therrien R, Richardson JB, Andersson M, Todman MG, Arden NK; DUROLANE Study Group. NASHA hyaluronic acid vs. methylprednisolone for knee osteoarthritis: a prospective, multi-centre, randomized, non-inferiority trial. Osteoarthritis Cartilage. 2014 Jan;22(1):17-25. doi: 10.1016/j.joca.2013.10.009. Epub 2013 Nov 1. PMID 24185114